CLINICAL TRIAL: NCT01209949
Title: Assessment of Subjects' Efficacy and Experiences Using Adapalene BPO Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US10179
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2012-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adapalene 0.1% and Benzoyl Peroxide 2.5% gel (Other)
  Interventions: Drug: Adapalene 0.1% and Benzoyl Peroxide 2.5% gel

INTERVENTIONS:
Drug: Adapalene 0.1% and Benzoyl Peroxide 2.5% gel — Apply adapalene BPO gel once daily in the evening for 12 weeks
  Other Names: Epiduo® Gel

SUMMARY:
The purpose of this study is to assess subjects' experiences using Adapalene BPO gel to treat mild to moderate acne vulgaris using efficacy measurements, quality of life instruments, and video diaries.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 16 to 25 years inclusive;
* Subjects with mild or moderate facial acne (Investigator's Global Assessment (IGA) = 2 or 3;
* A minimum of 10 inflammatory lesions (papules and pustules) on the face (excluding the nose);
* Subjects who agree to be photographed at each visit;
* Subjects who agree to be video recorded by study designated staff members. They should be able to clearly and comfortably communicate their responses to questions and express their thoughts related to their disease and treatment throughout the study

Exclusion Criteria:

* Subjects with nodules, cysts, acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.) or severe acne requiring systemic treatment;
* Subjects with a wash-out period for topical acne treatment on the face less than 30 days
* Subjects with a wash-out period for systemic acne treatment less than 30 days with the exception of isotretinoin which requires a washout of 4 months;
* Subjects who are currently being treated with antibiotics;
* Subjects who foresee intensive ultraviolet (UV) exposure during the study (mountain sports, UV radiation, sunbathing, tanning beds, etc.);
* Subjects who refuse photographic and videography procedures and/or refuse to sign a full release for their use in promotional materials

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Thomas J. Stephens and Associates, Carrollton, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on October 7, 2010 and the last subject was enrolled on October 12, 2010.
  Types of location: Investigative site was located at a research center.
Pre-assignment Details: Wash-out period up to baseline was 30 days for topical and systemic acne treatments with the exception of isotretinoin, which had a wash-out period of 4 months.
Groups:
- Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel: Adapalene 0.1% and Benzoyl Peroxide 2.5% gel - apply topically to the face once daily in the evening for 12 weeks
Period: Overall Study
Arm/Group | Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.5 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were a Success (Subject's Global Assessment of 'Clear' or 'Almost Clear') at Week 12
Description: Number of participants who were a Success (Subject's Global Assessment of 'Clear or 'Almost Clear') at week 12. Subject's Global Assessment is measured on a scale (Clear, Almost Clear, Mild, Moderate, Severe, Very Severe) with Clear being best and Very Severe being worst.
Time Frame: 12 weeks
Population: Modified ITT (subjects with a baseline and week 12 visit)
Measure: Number; unit: participants
Arm/Group | Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel
Number analyzed (Participants) | 27
participants | 18

2. Secondary Outcome: Percent Change From Baseline in Lesion Counts (Inflammatory, Non-inflammatory, and Total) at Week 12.
Description: Mean percent change from baseline in lesions counts (inflammatory, non-inflammatory, and total) at week 12.
Time Frame: Week 12
Population: Modified ITT (subjects with a baseline and week 12 visit)
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel
Number analyzed (Participants) | 27
percent change from baseline
  Inflammatory Lesions | -44.1 (34.79)
  Noninflammatory Lesions | -57.1 (19.83)
  Total Lesions | -49.7 (24.06)

3. Secondary Outcome: Number of Participants With Tolerability Assessments Resulting in an Adverse Event
Description: Number of participants with tolerability assessments resulting in an adverse event. Tolerability assessments include erythema (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe); Scaling (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe); Dryness (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe); Stinging/Burning (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) with a score of None being best and a score of Severe being worst.
Time Frame: 12 weeks
Population: Safety
Measure: Number; unit: participants
Arm/Group | Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel
Number analyzed (Participants) | 30
participants | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Adapalene 0.1% and Benzoyl Peroxide 2.5% Gel
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.